CLINICAL TRIAL: NCT05602649
Title: The Impact of Product Formulation on the Pharmacokinetics and Pharmacodynamics of Cannabis Edibles
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00354926; 1R01DA057201-01 (NIH)
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Cannabis Use
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions in a randomized order.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Placebo Gummy (Placebo Comparator): Participants will self-administer a gummy containing 0mg THC
  Interventions: Drug: Placebo
- Low Dose Gummy (Experimental): Participants will self-administer a gummy containing 10mg THC
  Interventions: Drug: Cannabis
- High Dose Gummy (Experimental): Participants will self-administer a gummy containing 25mg THC
  Interventions: Drug: Cannabis
- Placebo Chocolate (Placebo Comparator): Participants will self-administer chocolate containing 0mg THC
  Interventions: Drug: Placebo
- Low Dose Chocolate (Experimental): Participants will self-administer chocolate containing 10mg THC
  Interventions: Drug: Cannabis
- High Dose Chocolate (Experimental): Participants will self-administer chocolate containing 25mg THC
  Interventions: Drug: Cannabis
- Placebo Beverage (Placebo Comparator): Participants will self-administer a beverage containing 0mg THC
  Interventions: Drug: Placebo
- Low Dose Beverage (Experimental): Participants will self-administer a beverage containing 10mg THC
  Interventions: Drug: Cannabis
- High Dose Beverage (Experimental): Participants will self-administer a beverage containing 25mg THC
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Cannabis will be orally ingested
  Other Names: marijuana
  Arms: High Dose Beverage; High Dose Chocolate; High Dose Gummy; Low Dose Beverage; Low Dose Chocolate; Low Dose Gummy
Drug: Placebo — Placebo will be orally ingested
  Arms: Placebo Beverage; Placebo Chocolate; Placebo Gummy

SUMMARY:
This study will examine the pharmacokinetics and pharmacodynamics of delta-9-tetrahydrocannabinol (THC)-infused chocolates, gummies, and drinks. Healthy adults (N=40) will complete 9 drug administration sessions, including an overnight stay prior to each session. Participants will consume THC containing products in a fasted state; following drug administration, the participants will complete cognitive and psychomotor tasks, subjective assessments, have blood collected, and vital signs monitored.

DETAILED DESCRIPTION:
The purpose of this study is to examine the pharmacokinetics (PK) and pharmacodynamics (PD) of 3 popular types of cannabis edibles: THC-infused chocolates, gummies, and drinks. This study will utilize a rigorous double-blind, placebo-controlled, within-subjects design. Healthy adults (N=40; 20 males, 20 females) will complete 9 outpatient drug administration sessions in a randomized order. After 8 hours of monitored fasting, participants will consume 1 of 3 types of edibles (chocolates, gummies, or drinks) that are representative of current retail cannabis products. Products will contain 0 (placebo), 10, or 25mg THC. PD assessments include a battery of cognitive/psychomotor performance tasks shown to be sensitive to oral cannabis at these doses and subjective drug effects. Blood samples will be drawn to measure THC and its primary metabolites. Vital signs will be recorded. These procedures will be completed during each of the 9 study sessions.

ELIGIBILITY:
Inclusion Criteria

* Have provided written informed consent.
* Be between the ages of 21 and 55.
* Be in good general health based on screening procedures (e.g., physical exam, medical history interview, vital signs, routine blood tests).
* Test negative for illicit drugs (including cannabis) and test negative for alcohol (0% BAC) at screening and before any study sessions.
* Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at admission for each session.
* Have prior experience using THC-dominant cannabis.
* Have a body mass index (BMI) in the range of 16 to 38 kg/m2.
* Have not donated blood in the past 30 days.

Exclusion Criteria

* Self-reported use of illicit drugs (e.g., amphetamine, cannabis, cocaine, methamphetamine, MDMA, LSD, ketamine, heroin, psilocybin, prescription medications not prescribed to the person) in the past 30 days.
* History of significant allergic reaction or significant hypersensitivity to cannabis or to any of the other ingredients in the study products.
* Current concomitant medication use that may interact with the study drug including inhibitors and inducers of CYP2CP and CYP3A4 as well as highly-protein bound drugs and drugs with a narrow therapeutic index such as warfarin, cyclosporine, and amphotericin B.
* History of or current evidence of a significant medical condition that, in the opinion of the investigator or medical staff, will impact the participant's safety or interfere with study outcomes.
* Evidence of current psychiatric condition (based on MINI for DSM-5).
* Been in treatment previously for cannabis use disorder.
* Receiving of any drug as part of a research study within the past 30 days.
* History of epilepsy or other serious medical condition.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Working memory performance as assessed by the Correct Trials on Paced Auditory Serial Addition Task (PASAT) | 8 hours
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. Total correct trials out of 90 recorded is primary outcome (lower scores indicate worse performance).
Psychomotor performance as assessed by the Correct Trials on the Digit Symbol Substitution Task(DSST) | 8 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Total correct trials in 90 seconds is primary outcome (lower scores indicate worse performance).
Attention as assessed by the Mean Distance from the Center Target Stimulus on the Divided Attention Task (DAT) | 8 hours
  Computerized version of the Divided Attention Task will be administered to assess attention. Mean distance (in computer pixels) of the mouse cursor from the center target stimulus is primary outcome (lower scores indicate worse performance).
Executive functioning as assessed by the Mean Distance from the Center Target Stimulus on the Divided Attention Task (DAT) | 8 hours
  Computerized version of the Divided Attention Task will be administered to assess executive functioning. Mean distance (in computer pixels) of the mouse cursor from the center target stimulus is primary outcome (lower scores indicate worse performance).
DRiving Under the Influence of Drugs (DRUID) application global impairment score - Acute cognitive impairment | 8 hours
  Acute cognitive impairment will be assessed with global impairment score(range 0-100) on the DRUID app (higher scores indicate greater impairment).
DRUID application global impairment score - Acute behavioral impairment | 8 hours
  Acute behavioral impairment will be assessed with global impairment score(range 0-100) on the DRUID app (higher scores indicate greater impairment).
"Like Drug Effect" as assessed by the Drug Effect Questionnaire (DEQ) | 8 hours
  The DEQ will be used to obtain subjective ratings of "like drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
"Want to take again" as assessed by the Drug Effect Questionnaire | 8 hours
  The DEQ will be used to obtain subjective ratings of "want to take drug again". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
CMax for THC | 8 hours
  Blood concentrations of THC will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentrations (Cmax) is determined as the highest concentration reached for each individual.
AUC for THC | 8 hours
  Blood concentrations of THC will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.

SECONDARY OUTCOMES:
CMax for THC metabolite - 11-OH-THC | 8 hours
  Blood concentrations of 11-OH-THC will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentrations (Cmax) is determined as the highest concentration reached for each individual.
CMax for THC metabolite- THCCOOH | 8 hours
  Blood concentrations of THCCOOH will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentrations (Cmax) is determined as the highest concentration reached for each individual.
AUC for THC metabolite - 11-OH-THC | 8 hours
  Blood concentrations of 11-OH-THC will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
AUC for THC metabolite - THCCOOH | 8 hours
  Blood concentrations of THCCOOH will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
Tmax for THC | 8 hours
  Blood concentrations of THC will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. Time to max concentration (Tmax) will be calculated for each cannabinoid.
Tmax for THC metabolite - 11-OH-THC | 8 hours
  Blood concentrations of 11-OH-THC will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. Time to max concentration (Tmax) will be calculated for each cannabinoid.
Tmax for THC metabolite - THCCOOH | 8 hours
  Blood concentrations of THCCOOH will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. Time to max concentration (Tmax) will be calculated for each cannabinoid.
Cmax for CBD | 8 hours
  Blood concentrations of CBD will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentrations (Cmax) is determined as the highest concentration reached for each individual.
Cmax for CBN | 8 hours
  Blood concentrations of CBN will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentrations (Cmax) is determined as the highest concentration reached for each individual.
Cmax for CBG | 8 hours
  Blood concentrations of CBG will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The maximum concentrations (Cmax) is determined as the highest concentration reached for each individual.
AUC for CBD | 8 hours
  Blood concentrations of CBD will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
AUC for CBN | 8 hours
  Blood concentrations of CBN will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
AUC for CBG | 8 hours
  Blood concentrations of CBG will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. The area under the curve (AUC) is calculated across all timepoints, minus the baseline.
Tmax for CBD | 8 hours
  Blood concentrations of CBD will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. Time to max concentration (Tmax) will be calculated for each cannabinoid.
Tmax for CBN | 8 hours
  Blood concentrations of CBN will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. Time to max concentration (Tmax) will be calculated for each cannabinoid.
Tmax for CBG | 8 hours
  Blood concentrations of CBG will be measured using quantitative liquid chromatography-tandem mass spectrometry (LC-MS-MS) analysis. Time to max concentration (Tmax) will be calculated for each cannabinoid.
Psychomotor performance as assessed by attempted Trials on the Digit Symbol Substitution Task(DSST) | 8 hours
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Number of attempted trials is a secondary outcome.
Working memory performance as assessed by Reaction Time on Paced Auditory Serial Addition Task (PASAT) | 8 hours
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. The secondary outcome is the mean reaction time (in milliseconds) to select correct responses.
Attention as assessed by the Number of peripheral integers correct on Divided Attention Task (DAT) | 8 hours
  Computerized version of the Divided Attention Task will be administered to assess attention. The secondary outcome is the number of peripheral stimuli correctly identified.
Executive functioning as assessed by the Number of peripheral integers correct on Divided Attention Task (DAT) | 8 hours
  Computerized version of the Divided Attention Task will be administered to assess executive functioning. The secondary outcome is the number of peripheral stimuli correctly identified.
"Unpleasant Drug Effect" as assessed by the Drug Effect Questionnaire | 8 hours
  The DEQ will be used to obtain subjective ratings of "unpleasant drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
"Feel Drug Effect" as assessed by the Drug Effect Questionnaire- | 8 hours
  The DEQ will be used to obtain subjective ratings of "feel drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.

CONTACTS AND LOCATIONS:
Overall Officials: Tory Spindle, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No